CLINICAL TRIAL: NCT04616664
Title: Diagnostic Accuracy of the "LLIFT", a Novel Non-invasive Biomarker for the Diagnosis of Non Alcoholic Fatty Liver (NAFL) and SteatoHepatitis (NASH) in a Population With High Risk of Metabolic Syndrome"
Acronym: LLIFT
Status: Completed | Type: Observational
Sponsor: University Hospital, Lille (Other)
Collaborators: RHU PreciNASH Task 1.4 (Unknown); Région Nord-Pas de Calais, France (Other)
Responsible Party: Sponsor
Other Study IDs: 2019_45; 2020-A01991-38 (Other: ID-RCB number,ANSM)
Record Dates: First submitted 2020-10-06; First posted 2020-11-05 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Obesity; NASH - Nonalcoholic Steatohepatitis
Keywords: NAFL; NASH screening; metabolic syndrome; Diagnostic Biomarker; non-invasive biomarker
MeSH Terms: conditions — Obesity; Non-alcoholic Fatty Liver Disease; Metabolic Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The NAFLD is the first cause of liver disease worldwide. The severe form of NAFLD, the NASH progresses to cirrhosis and is responsible of liver mortality. The diagnosis of NASH requires liver biopsy that cannot be used for the screening of the disease.

The broad prevalence of the disease limits also the generalization of liver biopsy even for diagnosis. There is an urgent need for the use and the validation of liver diagnosis biomarkers for the diagnosis of NASH.

ELIGIBILITY:
Inclusion Criteria:

* Patients with 1 at least of the following metabolic criteria :

  * BMI > 30 kg/m²,
  * Type 2 diabetes (glycemia > 1.26 g/L or under therapy)
  * hypertension (> 140 mmHg / 90 mmHg or under therapy) associated with increased hepatic enzymes
* Indication of NAFLD evaluation
* Patients written consent
* Affiliated to a social insurance

Exclusion Criteria:

* Contraindications for liver biopsy or MRI.
* Other confounding cause of liver disease (HCV, HBV, HCC, autoimmune liver disease, Hemochromatosis, Wilson disease.
* alcohol consumption higher than 140g/week for women and 210g/week for men
* Previous history of alcohol abuse (addiction).
* Eluding stent < 6 month or acute coronary syndrome within 1 year or non-eluding stent within 6 weeks.
* Hepatocellular carcinoma
* Being processed Cancer (chemotherapy, radiotherapy or hormone therapy)
* Pregnant or breastfeeding women.
* Drug abuse within the past year.
* Mentally unbalanced patients, under supervision or guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients are followed in the cardiology, endocrinology, hepatology, hepatologic surgery and bariatric surgery units of the CHU de Lille and regional centers and presente type 2 diabetes or blood pressure hypertension associated with increased hepatic enzyme.
  Patients will be referred to the hepatology units and included in the study
Sampling Method: Probability Sample
Enrollment: 158 (Actual)
Dates: Start 2021-02-16 (Actual); Primary Completion 2024-01-17 (Actual); Study Completion 2024-01-17 (Actual)

PRIMARY OUTCOMES:
The Area under receiver operating characteristic (ROC) curve (AUC) of the LLIFT (Lille LIver Fat Test)-NASH score | Baseline
  The variables constituting the calculation algorithm are : clinical data (age, gender, BMI, diabetes status), biological data (AST, ALT, GCT, fasting glucose, HbA1c, triglyceride,...) and genetic polymorphism

SECONDARY OUTCOMES:
The Area under receiver operating characteristic (ROC) curve (AUC) of the LLIFT (Lille LIver Fat Test)- steatosis score | Baseline
  The variables constituting the algorithm are : clinical data (age, gender, BMI, diabetes status), biological data (AST, ALT, GCT, fasting glucose, HbA1c, triglyceride,..), genetic polymorphism.
Assessment of the correlation between the LLIFT score and the NAS score | Baseline
  The NAS score is a stratification based on steatosis, ballooning and lobular inflammation.

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume Lassailly, MD, Principal Investigator — University Hospital, Lille
Locations (7):
- France (7):
  - Chu Amiens Picardie, Amiens
  - CH ARRAS, Arras
  - CH de Douai, Douai
  - CH LENS, Lens
  - Hop Claude Huriez Chu Lille, Lille
  - GHIRCL saint Philibert, Lomme
  - Ch Valenciennes, Valenciennes